CLINICAL TRIAL: NCT02348190
Title: Fat Induced Insulin Resistance and Atherosclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 4148
Record Dates: First submitted 2015-01-22; First posted 2015-01-28 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Other Fatty Acid Oxidation Disorders; Diabetes Mellitus; Insulin Resistance
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — Lipids; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lipid/heparin (Active Comparator): 16 healthy volunteers will undergo euglycemic - hyperinsulinemic clamping without radioactive isotopes and with (n=16) lipid/heparin co-infusion for 8 hours.
  Interventions: Other: Lipid/heparin
- Control (Placebo Comparator): 16 healthy volunteers will undergo euglycemic - hyperinsulinemic clamping without radioactive isotopes and without (n=16) lipid/heparin co-infusion for 8 hours.
  Interventions: Other: Lipid/heparin

INTERVENTIONS:
Other: Lipid/heparin — 32 healthy volunteers will undergo euglycemic - hyperinsulinemic clamping without radioactive isotopes and with (n=16) and without (n=16) lipid/heparin co-infusion for 8 hours.
  Serial (at 0, 1, 2 and 4 h) muscle and fat biopsies and serial blood samples (q' 1 h) will be obtained. The following measurements will be obtained in muscle biopsies and T-cell extracts: PKC-βI and II and PKC-δ, IKK, IκB-α, NFκB, IRS-1 tyrosine phosphorylation, IRS-1 associated PI3- kinase, ICAM, VCAM and e-selectin mRNAs.

SUMMARY:
The overall objective of the current proposal is to strengthen the putative link between FFA induced insulin resistance and atherosclerotic vascular disease (ASVD). To this end, the investigators will test the following hypotheses: 1) that FFA induced activation of protein kinase C βII (PKC β II) and δ and other serine kinases such as IκB kinase (IKK) in human muscle is associated with a decrease in insulin stimulated tyrosine phosphorylation of the insulin receptor substrate-1 (IRS-1) and of IRS-1 associated phosphatidylinositol 3 (PI3) kinase; 2) that these changes precede the development of insulin resistance; 3) that the decrease in IκB-α results in activation of nuclear factor κB (NFκB) and the expression of adhesion molecules and cytokines; 4) that PKC and IKK are involved in producing insulin resistance and activation of the IκB/ NFκB pathway and lastly 5) that the same mechanisms operative in healthy volunteers are also operative in patients with T2DM.The investigators will test these hypotheses in normal (current) and diabetic volunteers (previously completed) . Euglycemic-hyperinsulinemic clamps will be performed with and without co-infusion of lipid plus heparin (to raise FFAs) and by obtaining serial muscle and fat biopsies and blood samples will be obtained for measurement of substrates, hormones, enzymes and metabolites.

DETAILED DESCRIPTION:
All subjects will be admitted to the GCRC in the afternoon before the tests (Day 1) and will undergo a thorough physical examination. Routine admission lab tests (including a 2-h 75g OGTT) and body composition measurements will be obtained. A standardized dinner will be served at ~ 6PM. The next (Day 2) after an overnight fast, IV lines will be placed (arms will be wrapped with a heating blanket and kept at 70ºF to arterialize venous blood).

The following studies will be performed.

Thirty-two healthy volunteers will undergo euglycemic - hyperinsulinemic clamping without radioactive isotopes and with (n=16) and without (n=16) lipid/heparin co-infusion for 8 hours.

Serial (at 0, 1, 2 and 4 h) muscle and fat biopsies and serial blood samples (q' 1 h) will be obtained. The following measurements will be obtained in muscle biopsies and T-cell extracts: PKC-βI and II and PKC-δ, IKK, IκB-α, NFκB, IRS-1 tyrosine phosphorylation, IRS-1 associated PI3- kinase, ICAM, VCAM and e-selectin mRNAs.

ELIGIBILITY:
Inclusion Criteria:

* The investigators plan to study 32 healthy normal subjects.
* These volunteers will be male and female, between the ages of 30 and 75 years and of all races.
* None of these volunteers will have a family history of diabetes or any other endocrine disorder and none will be taking any medications.

Exclusion Criteria:

* Patients with chronic health problems including cardiovascular, pulmonary, hematologic (*Hb< 9 g/dl), renal (serum creatinine > 1.8 mg/dl), hepatic disease, AIDS or other chronic infectious disease will be excluded.
* Pregnant women will be excluded. Non-pregnant women will be studied during the follicular phase of their menstrual cycle. If needed, a pregnancy test will be performed to exclude pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2003-06; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
protein kinase C enzyme activity in tissue samples | baseline, 1 hour, 2 hour, 4 hours
  The following measurements will be obtained in muscle biopsies: PKC-βI and II and PKC-δ, IKK, IκB-α, NFκB, IRS-1 tyrosine phosphorylation, IRS-1 associated PI3- kinase, ICAM, VCAM and e-selectin mRNAs.

SECONDARY OUTCOMES:
Insulin sensitivity | 0, 1, 2, 3, 4, 5, 6, 7, 8 hours
  Glucose infusion rates during the 8 hour euglycemic-hyperinsulemic clamp will be calculated.
Free fatty acids | 0, 1 2, 3, 4, 5, 6, 7 ,8 hours
  Free fatty acid levels will be measured by standard methods in the investigator's laboratory
protein kinase C enzyme activity in T cells | 0, 1, 2, 3, 4, 5, 6, 7, 8 hours
  T cell extracts will be used to assay PKC, IKK, IκB-α, NFκB and VCAM, ICAM and e-selectin mRNA.

CONTACTS AND LOCATIONS:
Overall Officials: Guenther Boden, MD, Principal Investigator — Temple University
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States